CLINICAL TRIAL: NCT05710315
Title: Single-center, Proof of Concept, Prospective Study Evaluating the Utility of RELiZORB™ for the Treatment of Feeding Intolerance in Critically Ill Adults With Multi-Organ Failure
Brief Title: Evaluating the Utility of RELiZORB™ for Treating Feeding Intolerance in Critically Ill Adults With Multi-Organ Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Alcresta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: INOVA-2023-42
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Multi Organ Failure; Exocrine Pancreatic Insufficiency
Keywords: Multi Organ Failure
MeSH Terms: conditions — Multiple Organ Failure; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Intervention Model Description: Two patients will receive enteral formula administered through RELiZORB™ as test subjects (will be excluded from analysis). Subsequently, patients will be randomized to RELiZORB™ vs placebo cartridges in a 1:1 ratio. Enteral nutrition will be administered through RELiZORB™ cartridges (up to 6 cartridges per day depending on the volume of enteral nutrition). Patients will be studied for a total of 5 days (considered to be the end of study). Patients will return to the original form of nutritional support per their routine clinical care.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RELiZORB (Experimental): RELiZORB™ cartridges connect in-line with existing enteral feeding pump tubing sets and patient extension sets or enteral feeding tubes.
  Interventions: Device: RELiZORB™
- Placebo (Placebo Comparator): Placebo cartridges connect in-line with existing enteral feeding pump tubing sets and patient extension sets or enteral feeding tubes
  Interventions: Other: Placebo

INTERVENTIONS:
Device: RELiZORB™ — RELiZORB cartridges will be used with routine enteral feedings for 5 days for randomized participants
  Arms: RELiZORB
Other: Placebo — Placebo cartridges will be used with routine enteral feedings for 5 days for randomized participants
  Arms: Placebo

SUMMARY:
The purpose of this research is to determine if the use of RELiZORB™ improves nutrition tolerance and helps critically ill patients meet their nutrition goals. RELiZORB™ is a digestive enzyme cartridge that contains lipase and works as a pancreatic enzyme replacement. It promotes breaking down fat and helps the body absorb it. The device connects with tube feedings to help the body with digestion.

RELiZORB™ is approved by the U.S. Food and Drug Administration (FDA) for use with tube feedings in patients 5 years of age or older. While the use of RELiZORB™ in this study is consistent with the FDA approval, the use of RELiZORB™ in patients with multi organ failure is not in the current standard of care practice at Inova Health Care facilities.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, parallel design study. A total of 32 adult patients who have been admitted to the Surgical or Medical Intensive Care Unit with evidence of MOF (defined as requiring mechanical ventilation and demonstrating at least one more system failure on the SOFA score on the day of ICU admission) and who have not yet been initiated on enteral nutrition or were initiated on enteral nutrition up to 48 hours prior.

After informed consent has been obtained, two patients will receive enteral formula administered through RELiZORB™ as test subjects (will be excluded from analysis). Subsequently, patients will be randomized to RELiZORB™ vs placebo cartridges in a 1:1 ratio. Enteral nutrition will be administered through RELiZORB™ cartridges (up to 6 cartridges per day depending on the volume of enteral nutrition). Patients will be studied for a total of 5 days (considered to be the end of study). Patients will return to the original form of nutritional support per their routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 - 89 years of age.
* Patients who have Multi-Organ Failure (MOF) (defined as requiring mechanical ventilation and demonstrating at least one more system failure on the SOFA score on the day of ICU admission).
* Patients who have not yet been initiated on enteral nutrition, yet enteral nutritional support is needed, or patients who have been initiated on enteral nutrition within the previous 48 hours. Enteral nutrition support defined as support planned to be given via any route connected to the gastrointestinal system (i.e., the enteral route). This includes tube feeding using nasogastric, nasoduodenal, gastrostomy, jejunostomy tubes, or similar.
* Patients who lack the capacity to consent for themselves may be included upon receiving consent from their legally authorized representatives.

Exclusion Criteria:

* Pregnant women and prisoners.
* Hypotension is attributed to suspected or confirmed cardiogenic shock.
* Evidence of unresolved intestinal obstruction, ischemia, bleeding, perforation, fistulas or tract discontinuity, or other contraindication for enteral nutrition.
* Sepsis suspected or confirmed due to an abdominal source and enteral nutrition is contraindicated.
* C. Difficile or other gastrointestinal infection that may manifest with diarrhea.
* Use of pancreatic hormone stimulant or inhibitor (e.g. octreotide, pancreatic enzyme supplements) during or immediately prior to hospital admission.
* Any other reason that the treating or investigator team considers to be a contraindication to enteral nutrition.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of RELiZORB™ in Enteral Nutrition Tolerance in Critically Ill Adults with Multiple Organ Failure Over Five Days | Duration of intervention (5 days)
  Efficacy will be assessed by the total calories administered, expressed as the percentage of goal nutrition calories achieved daily, compared between the two groups over the five-day study period

SECONDARY OUTCOMES:
Number of intolerance-related enteral nutrition pauses | Duration of intervention (5 days)
  The number of unplanned enteral nutrition pauses due to enteral nutrition intolerance
Insulin units used | Duration of intervention (5 days)
  Insulin units used
Change in fecal elastase | From Baseline to end of intervention at 5 days
  Change in fecal elastase as a measure of clinical exocrine pancreatic insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: George Kasotakis, MD MPH, Principal Investigator — Inova Fairfax Medical Campus
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Background] Stevens J, Wyatt C, Brown P, Patel D, Grujic D, Freedman SD. Absorption and Safety With Sustained Use of RELiZORB Evaluation (ASSURE) Study in Patients With Cystic Fibrosis Receiving Enteral Feeding. J Pediatr Gastroenterol Nutr. 2018 Oct;67(4):527-532. doi: 10.1097/MPG.0000000000002110. PMID 30074573
- [Background] Freedman S, Orenstein D, Black P, Brown P, McCoy K, Stevens J, Grujic D, Clayton R. Increased Fat Absorption From Enteral Formula Through an In-line Digestive Cartridge in Patients With Cystic Fibrosis. J Pediatr Gastroenterol Nutr. 2017 Jul;65(1):97-101. doi: 10.1097/MPG.0000000000001617. PMID 28471913
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Wang S, Ma L, Zhuang Y, Jiang B, Zhang X. Screening and risk factors of exocrine pancreatic insufficiency in critically ill adult patients receiving enteral nutrition. Crit Care. 2013 Aug 7;17(4):R171. doi: 10.1186/cc12850. PMID 23924602
- [Background] Saberi F, Heyland D, Lam M, Rapson D, Jeejeebhoy K. Prevalence, incidence, and clinical resolution of insulin resistance in critically ill patients: an observational study. JPEN J Parenter Enteral Nutr. 2008 May-Jun;32(3):227-35. doi: 10.1177/0148607108316195. PMID 18443133
- [Background] Nordenstrom J, Carpentier YA, Askanazi J, Robin AP, Elwyn DH, Hensle TW, Kinney JM. Free fatty acid mobilization and oxidation during total parenteral nutrition in trauma and infection. Ann Surg. 1983 Dec;198(6):725-35. doi: 10.1097/00000658-198312000-00011. PMID 6416194
- [Background] Kutsogiannis J, Alberda C, Gramlich L, Cahill NE, Wang M, Day AG, Dhaliwal R, Heyland DK. Early use of supplemental parenteral nutrition in critically ill patients: results of an international multicenter observational study. Crit Care Med. 2011 Dec;39(12):2691-9. doi: 10.1097/CCM.0b013e3182282a83. PMID 21765355
- [Background] Kelly MK. Bedside caregivers as change agents: implementation of early enteral nutrition in critical care. Crit Care Nurs Clin North Am. 2014 Jun;26(2):263-75. doi: 10.1016/j.ccell.2014.02.001. PMID 24878211
- [Background] Jarden RJ, Sutton LJ. A practice change initiative to improve the provision of enteral nutrition to intensive care patients. Nurs Crit Care. 2015 Sep;20(5):242-55. doi: 10.1111/nicc.12107. Epub 2014 Jul 18. PMID 25040624
- [Background] Jordan EA, Moore SC. Enteral nutrition in critically ill adults: Literature review of protocols. Nurs Crit Care. 2020 Jan;25(1):24-30. doi: 10.1111/nicc.12475. Epub 2019 Oct 10. PMID 31602712
- [Background] Compton F, Bojarski C, Siegmund B, van der Giet M. Use of a nutrition support protocol to increase enteral nutrition delivery in critically ill patients. Am J Crit Care. 2014 Sep;23(5):396-403. doi: 10.4037/ajcc2014140. PMID 25179035
- [Background] Doig GS, Heighes PT, Simpson F, Sweetman EA, Davies AR. Early enteral nutrition, provided within 24 h of injury or intensive care unit admission, significantly reduces mortality in critically ill patients: a meta-analysis of randomised controlled trials. Intensive Care Med. 2009 Dec;35(12):2018-27. doi: 10.1007/s00134-009-1664-4. Epub 2009 Sep 24. PMID 19777207
- [Background] Marik PE, Zaloga GP. Early enteral nutrition in acutely ill patients: a systematic review. Crit Care Med. 2001 Dec;29(12):2264-70. doi: 10.1097/00003246-200112000-00005. PMID 11801821
- [Background] Tian F, Heighes PT, Allingstrup MJ, Doig GS. Early Enteral Nutrition Provided Within 24 Hours of ICU Admission: A Meta-Analysis of Randomized Controlled Trials. Crit Care Med. 2018 Jul;46(7):1049-1056. doi: 10.1097/CCM.0000000000003152. PMID 29629984
- [Background] Hejazi N, Mazloom Z, Zand F, Rezaianzadeh A, Amini A. Nutritional Assessment in Critically Ill Patients. Iran J Med Sci. 2016 May;41(3):171-9. PMID 27217600
- [Background] Elpern EH, Stutz L, Peterson S, Gurka DP, Skipper A. Outcomes associated with enteral tube feedings in a medical intensive care unit. Am J Crit Care. 2004 May;13(3):221-7. PMID 15149056
- [Background] Osooli F, Abbas S, Farsaei S, Adibi P. Identifying Critically Ill Patients at Risk of Malnutrition and Underfeeding: A Prospective Study at an Academic Hospital. Adv Pharm Bull. 2019 Jun;9(2):314-320. doi: 10.15171/apb.2019.037. Epub 2019 Jun 1. PMID 31380259
- [Background] Wray CJ, Mammen JM, Hasselgren PO. Catabolic response to stress and potential benefits of nutrition support. Nutrition. 2002 Nov-Dec;18(11-12):971-7. doi: 10.1016/s0899-9007(02)00985-1. PMID 12431720
- [Background] Lew CCH, Yandell R, Fraser RJL, Chua AP, Chong MFF, Miller M. Association Between Malnutrition and Clinical Outcomes in the Intensive Care Unit: A Systematic Review [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):744-758. doi: 10.1177/0148607115625638. Epub 2016 Feb 2. PMID 26838530